CLINICAL TRIAL: NCT02276339
Title: The Role of the Peroneus Brevis and Peroneus Longus in Patients With Chronic Ankle Instability and the Effect of an Exercise Intervention
Brief Title: Muscle Activation in Chronic Ankle Instability and the Effect of an Exercise Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Principal Investigator, Dr Ulrik McCarthy Persson, Director of Sports Physiotherapy Masters programme UCD, Lecturer and Research supervisor, University College Dublin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS-13-50-OShea-McCarthy
Record Dates: First submitted 2014-10-13; First posted 2014-10-28 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Ankle Injuries
MeSH Terms: conditions — Ankle Injuries | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm ankle exercise intervention (Experimental): Chronic Ankle Instability Group assessed pre and post a 6 week eccentric - concentric exercise intervention
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — The exercise intervention will consist of an individual home-based progressive eccentric-concentric strengthening programme. Patients will be reviewed every two weeks during their rehabilitation; exercises will be progressed accordingly by their physiotherapist.

SUMMARY:
This study aims to investigate the activity patterns of the peroneal muscle group, in individuals with a history of chronic ankle instability (CAI) of the ankle injuries compared with individuals without ankle problems. The study also aims to determine the effect of a targeted exercise programme on this muscle group in patients with CAI.

Research on this topic may provide important insight on the roles of these muscles in chronic ankle instability and investigate whether specific strengthening programmes are effective in this complex patient category.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the role of the peroneus brevis (PB) and peroneus longus (PL) muscles in patients with chronic ankle instability and to determine whether an eccentric- concentric focused training intervention has an effect on these muscles.

Volunteers will be recruited from Orthopaedic Clinics and the Musculoskeletal Assessment Clinics in St. Vincent's University Hospital. Posters and information leaflets will be supplied to areas where volunteers are being sought. A study information sheet will be given to the patient and written consent will be obtained prior to commencing the investigative study.

Inclusion Criteria The selection criteria for chronic ankle instability (CAI) patients will be based on the position statement of the International Ankle Consortium (Gribble et al. 2013).

* A history of at least 1 significant ankle sprain
* A history of the previously injured ankle joint "giving way", and/or recurrent sprain, and/or "feelings of instability". Self-reported ankle instability confirmed with validated ankle instability-specific questionnaire: The Cumberland Ankle Instability Tool (CAIT). CAIT is a simple, valid, and reliable tool to measure severity of functional ankle instability.
* A general self-reported foot and ankle function questionnaire is also completed. The Foot and Ankle Ability Measure (FAAM): The FAAM is a reliable, responsive, and valid measure of physical function for individuals with a broad range of musculoskeletal disorders of the lower leg, foot, and ankle.

Exclusion Criteria

* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function (ie, sprains, fractures), resulting in at least 1 interrupted day of desired physical activity
* Any Neurological problem that would affect muscle function of the lower limb
* Pregnant Women
* Participants under 18 and over 65 Controls
* Healthy Volunteers (Control) will be age and sex matched to their CAI variants
* Will have no previous history of significant ankle sprain, which interrupted desired physical activity.

CAI patients will then be referred on for two radiological examinations in St. Vincent's

Hospital to aid diagnosis:

1. A diagnostic ultrasound will be performed by Dr. Eric Heffernan to look at peroneal tendon pathology and ligament character (thickening and continuity).
2. Stress Fluoroscopy (Anterior Drawer and Talar Tilt) will be performed by Professor Robert Flavin to assess for biplanar instability and to out rule subtalar instability.

Both participants with CAI and participants without ankle instability will undergo Surface electromyography (S-EMG) assessment of the PL, PB and Tibialis Anterior (TA) in both static and dynamic conditions in the University College Dublin School of Public Health, Physiotherapy & Population science (SPHPPS) motion analysis laboratory (This assessment process will initially be piloted on a healthy volunteer) Muscle onset will be determined and S-EMG will also normalized to Max Voluntary Contraction (MVC) determining the magnitude of activation, during Single leg Stance, wobble-board standing, walking, calf-raise exercise, tip-toe walking, jogging and a jump-landing task.

Kinematic variables (degrees of movement and speed) will also be re-coded using CODA motion capture system during the movement tasks.

The participants will be performing the functional tests on a force platform to allow for assessment of kinetic variables measuring ground reaction force and measures of postural control.

Following S-EMG testing the CAI subjects will commence a six-week eccentric-concentric focused exercise programme.

The exercise intervention will consist of an individual home-based progressive eccentric-concentric strengthening programme. Patients will be reviewed every two weeks during their rehabilitation; exercises will be progressed accordingly by their physiotherapist.

Patients will be supplied with exercise diaries to assist with adherence to the exercise protocol.

At the end of the six-week programme they will undergo repeat S-EMG testing and complete the self-reported ankle questionnaires used at pre-test phase.

If using a power level of 80% and 5% significance, a sample size of 13 participants for each study group would be required for this study. To allow for a 23% dropout rate we will aim to recruit 16 patients to each group.

ELIGIBILITY:
Inclusion Criteria:

The selection criteria for CAI patients will be based on the position statement of the International Ankle Consortium (2013).

* A history of at least 1 significant ankle sprain
* A history of the previously injured ankle joint "giving way", and/or recurrent sprain, and/or "feelings of instability". Self-reported ankle instability confirmed with validated ankle instability-specific questionnaire: The Cumberland Ankle Instability Tool. CAIT is a simple, valid, and reliable tool to measure severity of functional ankle instability (Hiller et al., 2006).
* A general self-reported foot and ankle function questionnaire is also completed. The Foot and Ankle Ability Measure: The FAAM is a reliable, responsive, and valid measure of physical function for individuals with a broad range of musculoskeletal disorders of the lower leg, foot, and ankle (Carcia et al., 2008).

Exclusion Criteria:

* Acute injury to musculoskeletal structures of other joints of the lower extremity in the previous 3 months that impacted joint integrity and function (ie, sprains, fractures), resulting in at least 1 interrupted day of desired physical activity
* Any Neurological problem that would affect muscle function of the lower limb
* Pregnant Women
* Participants under 18 and over 65

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Surface EMG | Assessed on day one, prior to intervention and at week 7 to assess change from baseline in EMG following the six-week intervention. Results presented 6 months later post analyses.
  Both participants with CAI and participants without ankle instability will undergo S-EMG assessment of the peroneus longus, peroneus brevis and tibialis anterior in both static and dynamic conditions in a university motion analysis laboratory (This assessment process will initially be piloted on a healthy volunteer) Muscle onset will be determined and S-EMG will also normalised to Max Voluntary Contraction (MVC) determining the magnitude of activation, during Single leg Stance, wobble-board standing, Walking, Calf-raise exercise, Tip-toe walking, jogging and a jump-landing task. Change in EMG will be assessed at week 7 following the six-week intervention.

SECONDARY OUTCOMES:
The Cumberland Ankle Instability Tool (CAIT) | Assessed on day one, prior to intervention and at week 7 to assess change from baseline in CAIT following the six-week intervention. Results presented 6 months later post analyses.
  CAIT is a simple, valid, and reliable tool to measure severity of functional ankle instability (Hiller et al., 2006).Change in CAIT will be assessed at week 7 following the six-week intervention.
The Foot and Ankle Ability Measure (FAAM) | Assessed on day one, prior to intervention and at week 7 to assess change from baseline in FAAM following the six-week intervention. Results presented 6 months later post analyses.
  The FAAM is a reliable, responsive, and valid measure of physical function for individuals with a broad range of musculoskeletal disorders of the lower leg, foot, and ankle (Carcia et al., 2008).Change in FAAM will be assessed at week 7 following the six-week intervention.
Patient global impression of change (PGIC) scale | Assessed at one time point only directly following the six-week intervention. Results presented 6 months later post analyses.
  Global rating of change (GRC) scales are very commonly used in clinical research, particularly in the musculo-skeletal area. These scales are designed to quantify a patient's improvement or deterioration over time, usually either to determine the effect of an intervention or to chart the clinical course of a condition. PGIC will only be assessed at one time point on week 7 following the six-week intervention.
Range and speed of movement | Assessed on day one, prior to intervention and at week 7 to assess change from baseline in movement following the six-week intervention. Results presented 6 months later post analyses.
  Kinematic variables (degrees of movement and speed) will also be recorded using CODA motion capture system during the movement tasks. Change in range and speed movement will be assessed at week 7 following the six-week intervention.
Kinetic measures of ground reaction force (GRF) | Assessed on day one, prior to intervention and at week 7 to assess change from baseline in GRF following the six-week intervention. Results presented 6 months later post analyses.
  The participants will be performing the functional tests on a force platform to allow for assessment of kinetic variables measuring ground reaction force and measures of postural control. Change in kinetic measures (GRF) will be assessed at week 7 following the six-week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ulrik McCarthy Persson, PhD, Study Director — University College Dublin
Locations (1):
- St. Vincent's University Hospital, Dublin, Leinster, Ireland

REFERENCES:
- [Background] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Background] Gribble PA, Delahunt E, Bleakley CM, Caulfield B, Docherty CL, Fong DT, Fourchet F, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino W, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Athl Train. 2014 Jan-Feb;49(1):121-7. doi: 10.4085/1062-6050-49.1.14. Epub 2013 Dec 30. PMID 24377963
- [Background] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343